CLINICAL TRIAL: NCT02908893
Title: Promoting Flu Vaccination Through a Mobile Wellness Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Evidation Health (Industry)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency); Army Research Office (ARO) (Unknown)
Responsible Party: Principal Investigator, Luca Foschini, Chief Data Scientist, Evidation Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EH-002
Record Dates: First submitted 2016-09-09; First posted 2016-09-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Not Condition-specific

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Salient (Experimental): Messages in the salient arm highlight the number of incentives (points) received by getting a flu shot and recording it through the wellness program app.
  Additionally, messages mention that flu shots can be received at the pharmacy while picking up an Rx.
  Users in the arm are matched up with a second user from the same arm, randomly. For each pair, the messages are sent to both users at the same time within the specified time window. Such time is picked to be the day in which the first user is most likely to pick up an Rx from a pharmacy.
  Interventions: Behavioral: In-app and push notification mobile messages
- NonSalient (Active Comparator): Messages in the non-salient arm highlight the benefits of getting vaccinated against flu, but make no mention of incentives received for getting vaccinated.
  Incentives would still be earned through the wellness program if the vaccination is recorded. Messages mention that flu shots can be received at the pharmacy while picking up an Rx.
  Users in the arm are matched up with a second user from the same arm, randomly. For each pair, the messages are sent to both users at the same time within the specified time window. Such time is picked to be the day in which the first user is most likely to pick up an Rx from a pharmacy
  Interventions: Behavioral: In-app and push notification mobile messages
- Control (No Intervention): Users in this group will not receive any message promoting flu vaccination. Incentives would still be earned through the wellness program if the vaccination is recorded.

INTERVENTIONS:
Behavioral: In-app and push notification mobile messages — Short messages (100-250 characters) are to be delivered to a mobile app both by push notification (i.e., appearing on the phone dashboard like a text message if the user has allowed notifications from the app) and in-app messages (visible in the news feed of the wellness program app when the app is opened). Messages contain a short title (30 characters) and 2-3 lines of text in the body (30 characters each).
  Arms: NonSalient; Salient

SUMMARY:
The investigators design a 6-week messaging campaign aimed at promoting flu vaccination among fully insured members of a national payer that participate in a wellness program offered by the insurer through a mobile app. Outcomes measured will include uptake in flu vaccination rate as measured by the insurer and engagement with the campaign through the app.

The goal of the research is to assess the effectiveness of pervasive computing messaging in promoting preventative care treatments such as flu shots. An additional goal is that of quantifying the importance of emphasizing incentives to increase efficacy of the messages.

ELIGIBILITY:
Inclusion Criteria:

* belongs to fully insured population
* continuous health coverage between January 1, 2015 and June 1, 2016
* has downloaded and installed the wellness platform app

Exclusion Criteria:

* has declined the messaging from the platform

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77983 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Increase in vaccination rate vs control | Up to 1 week after the end of each of the three batches of the intervention (Oct 1/15/28 2016)
  Increase in vaccination rate of anyone messaged relative to the control condition
Increase in vaccination rate of salient vs non-salient | Up to 1 week after the end of each of the three batches of the intervention (Oct 1/15/28 2016)
  Increase in vaccination rate of those who received salient incentives messages vs those who received generic messages

SECONDARY OUTCOMES:
Decrease in medically attended flu events of messaged vs control | Up to 1 week after the end of each of the three batches of the intervention (Oct 1/15/28 2016)
  Decrease in observed flu rate for messaged users
Increase in reporting of flu vaccination through wellness app of salient vs non-salient | Up to 1 week after the end of each of the three batches of the intervention (Oct 1/15/28 2016)
  Increase in reporting vaccination through the wellness program app following messages
Increase in vaccination rate for users messaged within 2 days before of an expected rx pick-up. | Up to 1 week after the end of each of the three batches of the intervention (Oct 1/15/28 2016)
  Increase in vaccination rate of users messaged within 2 days before an expected Rx pick up from a pharmacy relative to their paired partners.
Increase in message open rate of Salient vs Non-salient arm | Up to 1 week after the end of each of the three batches of the intervention (Oct 1/15/28 2016)
  Increase in open rate of sent messages through the wellness program app of salient vs non salient arm

CONTACTS AND LOCATIONS:
Locations (1):
- Evidation Health, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated outcome data may be shared.

REFERENCES:
- [Derived] Lee WN, Stuck D, Konty K, Rivers C, Brown CR, Zbikowski SM, Foschini L. Large-scale influenza vaccination promotion on a mobile app platform: A randomized controlled trial. Vaccine. 2020 Apr 16;38(18):3508-3514. doi: 10.1016/j.vaccine.2019.11.053. Epub 2019 Nov 29. PMID 31787410